CLINICAL TRIAL: NCT02089282
Title: Clavicular Shortening Post-fracture - Does it Change? - a Prospective Study of 70 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-369
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Stability of Clavicular Fractures Within the First 3 Weeks
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clavicle fractures
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound

SUMMARY:
In an attempt to answer if clavicular length changes after a fracture e.g. that any shortening becomes worse or better, 70 patients will be followed 3 times over 21 days using a novel ultrasound method.

ELIGIBILITY:
Inclusion Criteria:

All patients who sustain a displaced medial, mid and lateral clavicle fracture from March 2014 to August 2015 referred from Slagelse and Holbæk emergency departments are eligible. The last patients are seen end of mid-July 2015 given the 21 days of follow up.

Exclusion Criteria:

Patients that have bilateral clavicle fractures and/or prior operations involving the clavicle are excluded. Malignant diagnoses are excluded.

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clavicular fractures
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in clavicular length | 3 weeks
  The dynamic testing of clavicular length and when or which fracures that are stabile.

SECONDARY OUTCOMES:
Oxford shoulder score | 21 days

OTHER OUTCOMES:
Constant score | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Holbæk sygehus, Holbæk, Vest-sjælland, Denmark